CLINICAL TRIAL: NCT00664729
Title: Diet, Exercise, Metabolism, and Obesity in Older Women:DEMO
Brief Title: Diet, Exercise, Metabolism, and Obesity in Older Women
Acronym: DEMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AG020583 (NIH); R01AG020583 (NIH)
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Abdominal Obesity; Metabolic Syndrome
Keywords: Abdominal; obesity; exercise; intensity; weight loss; women
MeSH Terms: conditions — Obesity, Abdominal; Metabolic Syndrome; Obesity; Motor Activity; Weight Loss | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Active Comparator): Caloric Restriction
  Interventions: Behavioral: Caloric Restriction
- 2 (Experimental): Caloric restriction + Moderate-intensity aerobic exercise
  Interventions: Behavioral: Caloric Restriction + Low-Intensity aerobic exercise
- 3 (Experimental): Caloric restriction + Vigorous-intensity aerobic exercise
  Interventions: Behavioral: Caloric Restriction plus High-intensity aerobic exercise

INTERVENTIONS:
Behavioral: Caloric Restriction — Reduced calorie diet (400 kcal/day deficit)
  Other Names: Diet Only
  Arms: 1
Behavioral: Caloric Restriction + Low-Intensity aerobic exercise — 400 kcal/day deficit plus 3 days/week aerobic exercise at 45-50% maximal aerobic fitness
  Other Names: Diet+Low-Intensity AEX
  Arms: 2
Behavioral: Caloric Restriction plus High-intensity aerobic exercise — 400 kcal/day deficit and 3 d/week of aerobic exercise at 65-75% maximal fitness
  Other Names: Diet+High-intensity AEX
  Arms: 3

SUMMARY:
Reductions in fat oxidation and resting metabolic rate (RMR) are associated with normal aging and are accelerated with menopause. As a result, postmenopausal women have an increased risk of abdominal obesity and ultimately the metabolic complications that lead to the insulin resistance syndrome and its associated risks (hyperlipidemia, type 2 diabetes, and coronary heart disease). Thus, there is a need to determine the most successful treatment to reduce visceral obesity in postmenopausal women. The purpose of this study is to determine if dietary-induced weight loss alone and/or weight loss combined with exercise at low and high- intensities differentially affect the reduction in visceral adipose tissue in postmenopausal women with abdominal obesity.

DETAILED DESCRIPTION:
Design Overview:

This study's protocol will last approximately 18 months. Phase 1 involves recruitment and screening followed by baseline research testing (Phase 2). Next, subjects will be randomly assigned to one of three 5-month treatments (Phase 3): diet and high-intensity exercise, diet and low-intensity exercise, or diet only. In the Maintenance Phase, subjects will return for visits at 6 & 12 months following the completion of their 5 month intervention.

Interventions:

All treatment groups will experience the same total weekly caloric deficit (-2800 kcal/wk), but will derive this deficit by different reductions in dietary intake and exercise energy expenditure. The weekly caloric deficit will be accomplished as follows: 1) the diet alone group will reduce dietary intake by ~2800 kcal/week (~400 kcal/day); 2) both exercise groups will expend ~400 kcal/wk in exercise energy expenditure and will reduce dietary intake by ~2400 kcal/wk (~340 kcal/day) to achieve the 2800 kcal/wk deficit.

The exercise will take place in an exercise facility at the Geriatric Research Center on the campus of the Wake Forest University/Baptist Medical Center. Two study personnel, including at least one trained technician, will supervise all exercise sessions. Emergency equipment will be kept on site during exercise sessions. Blood pressure and heart rate will be measured and recorded before each exercise session and participants will warm-up by walking for 3-5 min at a slow pace. Women will use the treadmill to exercise at an intensity of 45-50% (low-intensity AEX) or 70-75% (high-intensity AEX) of VO2max. Both groups will exercise 3 d/wk and duration of exercise will progress from 10-15 min the 1st week to 55 min by the end of the 6th week and thereafter for the low-intensity AEX group. The duration of exercise for the high-intensity AEX group will progress from 10-15 min the 1st week to 30 min by the end of the 6th week and thereafter. Injuries are minimized by a feasible progression of exercise duration as well as careful monitoring of proper footwear and stretching exercises.

The diet intervention will consist of monthly meetings with a registered dietitian along with consuming a hypocaloric diet provided by the GCRC metabolic kitchen. Subjects will be asked to pick up their food three times a week. Two meals per day will be provided. In addition, a calcium supplement (1000mg) will be provided. Subjects will be required to keep a diary of other foods consumed including the calcium supplement. The diets will be composed of 50-60% carbohydrate, 15-20% protein, and 25-30% fat with adequate amounts of essential nutrients. The number of calories given to each subject will be estimated from energy expenditure estimates in combination with an activity factor. The diet only group will be provided with an approximate 400 kcal/day energy deficit diet, while both exercise groups will be provided with an approximate 340 kcal/day energy deficit diet. Menus and specific food choices will be determined by GCRC dietitians in consultation with each research subject.

ELIGIBILITY:
Inclusion Criteria:

* Currently 50 - 70 years of age (at screening)
* Post-menopausal at least 1 year
* Waist diameter of at least 34"
* Able to attend exercise classes 3 times per week
* BMI between 25 & 40 kg/m2
* MMSE > 25

Exclusion Criteria:

* Exercises regularly (ie- more than twice a week for more than 15 minutes per session)?
* Uncontrolled diabetes mellitus or insulin-controlled diabetes?
* Does not drive and does not have a reliable way to pick up meals once a week
* Cancer in past 5 years except skin cancer
* Unwilling or unable to eat prepared foods (non-compliant during test week)
* Unwilling or unable to record food intake accurately
* Self-reported weight loss or gain >5% in past 6 months
* Smoking within past year, or use of tobacco or nicotine product
* Coronary artery disease, liver disease, renal disease, or other systemic disorders
* Pulmonary disease
* Current use of thiazide diuretics, beta blockers or steroids
* Current use of more than one anti-hypertensive medication
* Current use of anti-depressants or hormone replacement therapy
* Gross physical impairment
* Blindness or retinopathy
* Triglyceride level >400 mg/dl
* Anemia (Hct < 37%)
* Contraindication to exercise by ECG or GXT

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2002-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Abdominal visceral fat volume | Baseline, follow-up

SECONDARY OUTCOMES:
HDL cholesterol Triglyceride concentrations Glucose tolerance | Baseline and Follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Nicklas, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Result] You T, Murphy KM, Lyles MF, Demons JL, Lenchik L, Nicklas BJ. Addition of aerobic exercise to dietary weight loss preferentially reduces abdominal adipocyte size. Int J Obes (Lond). 2006 Aug;30(8):1211-6. doi: 10.1038/sj.ijo.0803245. Epub 2006 Jan 31. PMID 16446745
- [Result] You T, Yang R, Lyles MF, Gong D, Nicklas BJ. Abdominal adipose tissue cytokine gene expression: relationship to obesity and metabolic risk factors. Am J Physiol Endocrinol Metab. 2005 Apr;288(4):E741-7. doi: 10.1152/ajpendo.00419.2004. Epub 2004 Nov 23. PMID 15562250
- [Derived] Wang X, You T, Murphy K, Lyles MF, Nicklas BJ. Addition of Exercise Increases Plasma Adiponectin and Release from Adipose Tissue. Med Sci Sports Exerc. 2015 Nov;47(11):2450-5. doi: 10.1249/MSS.0000000000000670. PMID 25811948
- [Derived] You T, Disanzo BL, Wang X, Yang R, Gong D. Adipose tissue endocannabinoid system gene expression: depot differences and effects of diet and exercise. Lipids Health Dis. 2011 Oct 28;10:194. doi: 10.1186/1476-511X-10-194. PMID 22035053
- [Derived] Nicklas BJ, Wang X, You T, Lyles MF, Demons J, Easter L, Berry MJ, Lenchik L, Carr JJ. Effect of exercise intensity on abdominal fat loss during calorie restriction in overweight and obese postmenopausal women: a randomized, controlled trial. Am J Clin Nutr. 2009 Apr;89(4):1043-52. doi: 10.3945/ajcn.2008.26938. Epub 2009 Feb 11. PMID 19211823